CLINICAL TRIAL: NCT00500630
Title: Objective Evaluation of Shoulder Pathology and Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: HO 22/04
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2007-07-13 (Estimated); Status verified 2007-07

CONDITIONS: Glenohumeral Osteoarthritis; Rotator Cuff Disease

INTERVENTIONS:
Device: Body fixed 3D sensors

SUMMARY:
The goal of this study was to clinically validate a new device for the objective outcome evaluation of adult patients undergoing shoulder surgery for glenohumeral osteoarthritis and rotator cuff disease, using the activities of daily living described in the Simple Shoulder Test (SST) as a reference.

The study was set up as a clinical trial including patients over an observation period of one year and a control group of subjects. Clinical evaluations will be made at baseline, 3 months, 6 months and 1 year after surgery by two independent observers. Miniature sensors each containing three 3D gyroscopes and three 3D accelerometers will allow computing new kinematic scores. They will be compared to the regular SST, DASH, ASES and Constant scores.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* patients with a unilateral rotator cuff disease implying a transfixiant supraspinatus rupture of at least 1 cm2, as determined by Magnetic Resonance Imaging (MRI), or a unilateral glenohumeral osteoarthritis stage II or III according the radiologic criteria published by Koss
* informed and signed consent

Exclusion Criteria:

* Patients who had a previous shoulder surgery (open or arthroscopic)
* Patients who had a contralateral shoulder pathology

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte M Jolles, MD, MSc, Study Director — Centre Hospitalier Universitaire Vaudois - University of Lausanne
Locations (1):
- Hopital Orthopédique de la Suiss Romande, Lausanne, CH, Switzerland